CLINICAL TRIAL: NCT02043184
Title: Improving Adherence to Oral Cancer Agents and Self Care of Symptoms Using an IVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Given, University Distinguished Professor, Michigan State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01CA162401-01A1 (NIH); 1R01CA162401 (NIH)
Record Dates: First submitted 2014-01-20; First posted 2014-01-23 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Prostatic Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Melanoma; Leukemia
Keywords: Neoplasms; Medication Adherence; Administration, Oral; Symptom Assessment; Neurobehavioral Manifestations; Depression; Behavioral Symptoms; Utilization
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Melanoma; Leukemia; Neoplasms; Medication Adherence; Neurobehavioral Manifestations; Depression; Behavioral Symptoms; Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard Care 12 weeks (Active Comparator): Standard care. Standard supportive care and Toolkit given at 12 weeks.
  Interventions: Behavioral: Interactive Voice Response (IVR) Reminders
- Standard Care 8 wks, Daily IVR 4 wks (Experimental): Interactive Voice Response (IVR) Reminders Daily delivery for the last 4 weeks of the study.
  Interventions: Behavioral: Interactive Voice Response (IVR) Reminders
- Daily IVR 8 weeks (Experimental): Interactive Voice Response (IVR) Reminders daily for the first 8 weeks of the study.
  Interventions: Behavioral: Interactive Voice Response (IVR) Reminders
- Daily IVR 4 wk, Every other day IVR 4 wk (Experimental): Interactive Voice Response (IVR) Reminders daily for the first 4 weeks of the study and every other day for weeks 4-8.
  Interventions: Behavioral: Interactive Voice Response (IVR) Reminders

INTERVENTIONS:
Behavioral: Interactive Voice Response (IVR) Reminders — Reminders tailored to the oral cancer medication(s) the patients are receiving delivered by interactive voice response system with referral to a self-management guide when symptoms exceed thresholds.

SUMMARY:
Improving Adherence to Oral Cancer Agents and Self Care of Symptoms Using an IVR The goals of this study are to improve adherence to oral chemotherapeutic medications and self-management of symptoms among cancer patients. More than 40 oral agents currently are on the market with projections that in three years 30% of the cancer treatment agents will be delivered in oral form. As a result, patients must assume responsibility for taking medications and self-management of associated side effects.

This longitudinal randomized trial tests and compares 'two strategies' for improving patient adherence to their oral cancer medication prescriptions to standard care. Both strategies incorporate symptom management support using an interactive voice response system (IVR) for symptom assessment and a printed evidence-based Medication Management and Symptom Management Toolkit (Toolkit) with helpful strategies and information for symptom management.

We will collaborate with NCI Comprehensive Cancer Centers to recruit patients into this study. Recruiters will identify patients as they are prescribed oral cancer medications, present the study to the patient, and ask them to consent to be part of the study.

Study Aims Following are the Aims of the study.

1. Cancer patients assigned to the intervention will have greater adherence to their prescribed regimen: a) at week 4 (immediate effect), and b) at weeks 8 and 12 (sustained effect).
2. When compared with patients receiving weekly assessments only, patients receiving weekly assessments plus daily adherence reminders and printed symptom management strategies for 4 weeks will report: lower symptom severity during weeks 2-4 that will be sustained at weeks 5-8, and at 12 weeks.

Two exploratory aims are assessed:

1. To test how patient characteristics (age, sex, depression), dose variation, symptom severity, and concurrent infusion therapy moderate the impact of the novel intervention on adherence at 4, 8, and 12 weeks.
2. To test the impact of the novel intervention on dose alterations, emergency department visits and hospital admissions over the 12 weeks in order to support the translation of this system into oncology practices.

DETAILED DESCRIPTION:
Design and Methods A unique feature of this study is that assessments, reminders, and symptom management strategies will be delivered by an Interactive Voice Response system (IVR). This system has been tested in a previous trial and in a pilot study of medication adherence; it received high satisfaction ratings from patients.

All patients will complete intake (baseline), 4 week, 8 week, and 12 week interviews for symptom severity, depression, beliefs about oral agents, self-efficacy, and pill count. Following the intake interview a computerized procedure will randomize patients to one of two groups: experimental and control. Patients in both arms will receive 12 weekly assessments of adherence to their oral cancer medications and symptom severity delivered by the IVR.

In addition, patients in the experimental group will receive daily reminder calls for 4 weeks delivered by the IVR. At the end of week 4 patients will be offered the option to reduce calls to every other day, or continue with daily reminders for weeks 5-8. Reminder calls will be tailored to the cycle of each medication. Daily reminder calls include a question to determine if medication changes have occurred. If this occurs, reminder calls are stopped and/or adjusted to the revised prescription. Patients in the experimental group will be mailed a Toolkit. Patients who report symptoms above designated thresholds during a weekly assessment call will be referred to the Toolkit to assist with self-management.

The control group will not receive IVR reminder calls during the first 8 weeks. Control group patients, who report difficulty taking their cancer medications as prescribed, will be randomized following the 8 week interview to either receive 4 weeks of daily IVR reminder calls during weeks 9-12, or to continue in the control group. Patients randomized to receive daily IVR reminder calls will receive a Toolkit following randomization (and if during their weekly assessment calls they report symptoms above designated thresholds they will be referred to the Toolkit to assist with self-management). Patients randomized to continue in the control group will receive a Toolkit upon completion of the 12 week interview.

Medical records will be audited for oral cancer medication changes during the study period as well as adverse toxic events noted, and scripts written.

Implications & Impact This research will identify and explore the factors (symptom severity, medication complexity, patient characteristics) affecting adherence to oral cancer medications and how symptom management might improve levels of adherence. This will allow patients to engage in their care and potentially transform the safety and quality of cancer care for patients on oral cancer medications.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Newly prescribed one of the designated oral cancer medications for treatment of cancer
* ECOG score of 0,1,or 2 OR Karnofsky score of 50 or higher
* Patient of one of the participating National Cancer Institute comprehensive cancer centers
* Able to speak, read and understand English
* Able and willing to receive phone calls

Exclusion Criteria:

* Difficulty hearing on the telephone
* Limited or no access to a touch tone phone
* Cognitive deficits
* Hospice care at enrollment
* Those prescribed a hormonal therapy for cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2013-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Medication Adherence using pill count and self report | 8 weeks

SECONDARY OUTCOMES:
Medication Self-Efficacy using Horne Measure | 8 weeks
  this assesses the ability to believe that they can adhere
Symptom Burden is determining the overall number of symptoms on the given symptom tool | 8 weeks
  The Given Symptom assessment tool is used
Symptom Interference is the interference with daily activities | 8 weeks
  This is an adaptation of the Cleeland Interference scale
Depression using the full Clinical Screening for depression measure | 8 weeks
  we are using the CESD
Physical Function using the Physical Function Scale | 8 weeks
  We use the PROMIS physical function measure
Healthcare Utilization is the use of Emergency room and Hospital admissions | 8 weeks
  This captures the use during the 8 weeks and is Emergency room use and hospital admissions including length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Given, PhD, Principal Investigator — Michigan State University; Charles Given, PhD, Principal Investigator — Michigan State University
Locations (8):
- United States (8):
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - MSU Breslin Cancer Center, Lansing, Michigan
  - Sparrow Cancer Center, Lansing, Michigan
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available.

REFERENCES:
- [Derived] Marshall VK, Given CW, Given BA, Lehto RH, Sikorskii A. Factors affecting medication beliefs among patients newly prescribed oral oncolytic agents. J Psychosoc Oncol. 2022;40(1):62-79. doi: 10.1080/07347332.2020.1855497. Epub 2020 Dec 11. PMID 33305993
- [Derived] Sikorskii A, Given CW, Given BA, Banik A, Krauss JC. Patient Engagement With an Automated Telephone Symptom Management Intervention: Predictors and Outcomes. Ann Behav Med. 2020 Jun 12;54(7):484-494. doi: 10.1093/abm/kaz067. PMID 31925414
- [Derived] Decker V, Sikorskii A, Given CW, Given BA, Vachon E, Krauss JC. Effects of depressive symptomatology on cancer-related symptoms during oral oncolytic treatment. Psychooncology. 2019 Jan;28(1):99-106. doi: 10.1002/pon.4916. Epub 2018 Oct 23. PMID 30311987